CLINICAL TRIAL: NCT02055079
Title: Pulsed Oral Sirolimus in Autosomal Dominant Polycystic Kidney Disease - The Vienna RAP Study
Brief Title: Pulsed Oral Sirolimus in Autosomal Dominant Polycystic Kidney Disease
Acronym: RAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Riegersperger, MD, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V5.1/20.1.2013; 2012-000550-60 (EudraCT Number); 15170 (Other Grant/Funding Number: Oesterreichische Nationalbank); 1060/2012 (Other: Ethics committee Medical University of Vienna)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Polycystic Kidney, Type 1 Autosomal Dominant Disease; Polycystic Kidney, Type 2 Autosomal Dominant Disease
Keywords: ADPKD; PKD; Polycystic kidney disease; Mammalian target of rapamycin; mTOR-I; Sirolimus
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases; Hereditary Sensory and Autonomic Neuropathies | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus (Experimental): Fixed oral dose of 3 mg Sirolimus (blinded) once weekly for 24 months.
  Interventions: Drug: Sirolimus
- Placebo (Placebo Comparator): Fixed oral dose of placebo (blinded) once weekly for 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Fixed oral dose of 3 mg sirolimus (blinded) once weekly for 24 months.
  Other Names: Rapamune
  Arms: Sirolimus
Drug: Placebo — Fixed oral dose of 3 mg placebo (blinded) once weekly for 24 months.
  Arms: Placebo

SUMMARY:
Sirolimus (SIR) has lead to a reduction of overall kidney size, a decrease in cyst density and general tubular cell proliferation in animal models, and to a reduction of the increase in creatinine and blood urea nitrogen by 34 and 39 percent respectively, as well as a reduction of cyst proliferation, expressed by a 30 percent reduction of overall kidney enlargement, a reduction in general cyst volume, and a reduction of the cyst volume density in the renal cortex in humans.

However, despite promising data from animal- and in vivo studies, most mammalian target of rapamycin inhibitor (mTOR-I) studies in patients with autosomal-dominant polycystic kidney disease (ADPKD) produced only subtle if any clinically relevant effects on cyst growth and the preservation of renal function.

In this study we will investigate if pulsed administration of SIR in a fixed weekly oral dose of 3 mg over 24 months compared to placebo significantly reduces cyst growth and preserves excretory renal function in patients with ADPKD and an estimated glomerular filtration (eGFR) rate below 60 mL/min per 1.73m2.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD, as confirmed by history, ultrasound, computed- or magnetic resonance tomography
* Eighteen years of age, or older
* Baseline eGFR below 60 mL/min per 1.73m2
* Negative serum pregnancy test prior to administration of sirolimus and agreement to use contraception throughout the study and three months after
* Written informed consent

Exclusion Criteria:

* Need for renal replacement therapy
* Pregnancy/lactation
* Plans to become pregnant in the near future
* Refusal to use sufficient contraception
* Proteinuria as defined as protein:creatinine ratio >1000 or >1g/d, respectively
* History of life threatening complications of ADPKD
* Evidence of active systemic- or localized major infection
* Evidence of infiltrate or consolidation on chest X-ray
* Use of any investigational drug or -treatment up to 4 weeks prior to enrolment and during the study
* Known allergy/hypersensitivity to sirolimus and its derivatives
* Medication that will interfere with the cytochrome P450 (CYP3A4/CYP3A5) system
* Total white blood cell count below or equal to 3000/mm3
* Platelet count below or equal to 100.000/mm3
* Fasting triglycerides above or equal to 400 mg/dL
* Fasting total cholesterol above or equal to 300 mg/dL
* Concomitant glomerular diseases
* Psychiatric disorders and any condition that might prevent full comprehension of the purposes and risks of the study
* History of malignancy, with the exception of adequately treated basal cell- and squamous cell carcinoma of the skin
* HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in kidney function from baseline to month 24 | Baseline, 24 months
  Fifty percent reduction in doubling of serum creatinine, or initiation of dialysis over a period of two years. Less or equal than 1.5 fold increase in serum creatinine without initiation of dialysis over two years is considered a beneficial outcome, increases in serum creatinine greater than 1.5 over two years or initiation of dialysis are considered a non-beneficial outcome.

SECONDARY OUTCOMES:
Change of safety parameters from baseline to month 24 | Baseline, 24 months
  Safety, change in proteinuria, as indicated by albumin/creatinine- and protein/creatinine ratio, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Riegersperger, MD, Principal Investigator — Medical University of Vienna; Gere Sunder-Plassmann, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Division of Nephrology and Dialysis, Department of Medicine III, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Riegersperger M, Herkner H, Sunder-Plassmann G. Pulsed oral sirolimus in advanced autosomal-dominant polycystic kidney disease (Vienna RAP Study): study protocol for a randomized controlled trial. Trials. 2015 Apr 23;16:182. doi: 10.1186/s13063-015-0692-3. PMID 25899445